CLINICAL TRIAL: NCT05314101
Title: TAS-102 Combined With Bevacizumab and Tislelizumab Third-line or Above in the Treatment of Liver Metastasis in Colorectal Cancer : An Open-label 、Phase Ⅱ Clinical Trial
Brief Title: TAS-102 Combined With Bevacizumab and Tislelizumab Third-line or Above in the Treatment of Liver Metastasis in Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBT001
Record Dates: First submitted 2022-03-19; First posted 2022-04-06 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-03

CONDITIONS: Immunotherapy; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Bevacizumab; trifluridine tipiracil drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TAS-102 combined with bevacizumab and tislelizumab (Experimental): TAS-102 combined with bevacizumab and tislelizumab third-line or above in the treatment of liver metastasis in colorectal cancer
  Interventions: Drug: Tislelizumab; Drug: bevacizumab; Drug: TAS-102

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks
Drug: bevacizumab — Participants will receive bevacizumab，5mg/kg，intravenously over 60 - 90 minutes, day 1 and day 15 of every 4 weeks
Drug: TAS-102 — Participants will receive TAS-102, 35mg/m2, bid，d1-d5, d8-d12 of every 4 weeks

SUMMARY:
To evaluate the clinical efficacy and safety of TAS-102 combined with bevacizumab and tislelizumab in third-line or above treatment in patients with advanced colorectal adenocarcinoma with liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients who provided informed consent and voluntarily enrolled
* Patients with liver metastasis of advanced colorectal adenocarcinoma with MSS confirmed by pathology;
* 18-75 years old;
* Measurable target lesions according to RECIST V1.1 assessment criteria;
* Progression after standard second-line treatment (irinotecan, oxaliplatin, or fluorouracil);
* 0 ~ 2 points according to ECOG quality of life score;
* Drugs can be taken orally
* Estimated survival ≥3 months;
* Women of childbearing age should comply with contraceptive measures if pregnancy test is negative;
* Ascites with no obvious symptoms and no clinical intervention;
* Adequate organ and bone marrow functions, ecg, blood, biochemical and other basic tests are not contraindications of chemotherapy;
* Adherence to scheduled visits, treatment plans, laboratory tests, and other study procedures Willingness and ability.

Exclusion Criteria:

* Previous application of TAS-102;
* Pregnant or lactating women;
* No contraception during the reproductive period;
* patients known to have a history of allergy to any study drug, similar drug or excipient;
* Patients with risk of massive gastrointestinal bleeding or gastrointestinal obstruction;
* Patients with a history of thromboembolism, except those caused by PICC;
* Patients with active infection;
* Patients with uncontrolled hypertension (systolic blood pressure ≥160 mmHg and diastolic blood pressure ≥90) MmHg);
* Patients with brain metastases with clinical symptoms or imaging evidence;
* Contraindications for treatment of other chronic diseases;
* Previous immunotherapy-related myocarditis, pneumonia, colitis, hepatitis, kidney Inflammation and other conditions, the current AE is still ≥2;
* According to THE NCI CTCAE 5.0 assessment criteria, there are all types of existing cases due to previous treatment Patients with grade ≥2 toxic reactions;
* Other conditions that the investigator determines are not suitable for inclusion in the study.
* Received any anti-tumor therapy and participated in other clinical studies within 4 weeks prior to enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 24 months
  Time from enrollment to the onset of disease progression or death.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | every 8 weeks (up to 24 months)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

OTHER OUTCOMES:
Overall survival (OS) | every 3 months (up to 24 months) ]
  Defined from date of Signing ICF to date of first documentation of death from any cause or censored at the date of the last follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- FujianCH, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No